CLINICAL TRIAL: NCT07038681
Title: Mediterranean Diet Intervention for Maternal Postpartum Cardiometabolic and Microbiome Health (MedMom Study): a Randomized Trial
Brief Title: Mediterranean Diet Intervention for Maternal Postpartum
Acronym: MedMom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MedMom
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Postpartum; Cardiometabolic Factors; Cardiac Reverse Remodeling
Keywords: Mediterranean Diet; Postpartum; Pregnancy; Cardiac Reverse Remodeling
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-treatment, one-period, parallel trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Hospital Dietary Care) (Placebo Comparator): Since all the pregnant women in this study have at least one of the following risk factors: obesity, diabetes or hypertension, nutritional follow-up is a standard-care procedure in the Portuguese National Health System, therefore the control group receive usual care from the nutritionist in the hospital.
  Interventions: Other: Control Group (Standard Hospital Dietary Care)
- Mediterranean Diet Intervention Group (Experimental): In addition to the standard-care follow-up in the Portuguese National Health System, the intervention group will have additionally three approaches within the intervention: i) one face-to-face appointment lasting 10 to 15 minutes conducted by a registered dietitian (3rd trimester: 30 - 35 gestational weeks); ii) a 13-page manual that accompanies the dietary education session, which is provided to each participant; and iii) five monthly newsletters sent via e-mail from two weeks after childbirth until the fifth month postpartum.
  Interventions: Other: Mediterranean Diet Intervention Group

INTERVENTIONS:
Other: Mediterranean Diet Intervention Group — In the same way as the control group, the intervention group receives standard nutritional care from the hospital nutritionist, since all the pregnant women have at least one of the following risk factors: obesity, diabetes or hypertension, nutritional - standard-care procedure in the Portuguese National Health System.
  Other Names: Diet group
  Arms: Mediterranean Diet Intervention Group
Other: Control Group (Standard Hospital Dietary Care) — The control group will receive standard care from the nutritionist in the hospital.
  Arms: Control Group (Standard Hospital Dietary Care)

SUMMARY:
The increasing prevalence of obesity during women's reproductive years highlights the need for effective strategies to improve nutritional literacy as a preventive approach to adverse postnatal outcomes.

This study outlines a protocol for a pilot randomized controlled trial assessing the potential of nutritional education sessions promoting the Mediterranean Diet (MedDiet) to improve adherence to this diet and evaluate its effects on cardiometabolic outcomes, namely on cardiac reverse remodeling, glycemic and blood pressure control, as well as on preconception weight recovery and changes in the fecal microbiota composition in pregnant women with obesity, hypertension, and/or diabetes.

Secondarily, this study aims to evaluate how this dietary intervention indirectly interferes with infants' exclusive breastfeeding and the introduction of complementary feeding. It includes a face-to-face session using an eye-catching 13-page manual, followed by five monthly newsletters sent by e-mail. Participants will be monitored at one, six, and twelve months postpartum to evaluate the intervention's effectiveness. Findings from this study will contribute to the development of an evidence-based nutritional education tool designed to improve maternal health outcomes, with potential applicability for both health professionals and pregnant and postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Adult female (>18 years old)
* Obesity
* Chronic arterial hypertension
* Type 2 diabetes
* Gestational hypertension
* Gestational diabetes

Exclusion Criteria:

* Preexisting cardiomyopathy;
* Renal disease;
* Chronic obstructive airway disease;
* Active systemic infection;
* Genetic syndromes;
* Type 1 Diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Mediterranean Diet Adherence | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum)
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the. Portuguese National Health System (Control Group: Standard Hospital Dietary Care)) on the percentage change of the Mediterranean Diet Adherence Screener (MEDAS) score.
  The MEDAS score ranges from 0 to 14, with higher scores indicating greater adherence to the Mediterranean Diet. Scores are commonly classified as follows:
  * Low adherence: < 7
  * Moderate adherence: 7-9
  * High adherence: ≥ 10

SECONDARY OUTCOMES:
Left Ventricular Reverse Remodeling Assessed by Echocardiography (Cardiac reserve remodeling) | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of dietary education counseling focused on Mediterranean Diet promotion (intervention group) vs control group on cardiac reverse remodeling, evaluated through echocardiographic measurements of cardiac structure and function during pregnancy and postpartum.
  Cardiac reverse remodeling will be assessed as the change (Δ) in left ventricular (LV) mass between the third trimester of pregnancy and 6 months postpartum.
  Conventional transthoracic echocardiography will be performed using a 3 MHz phased-array probe (ACUSON SC2000 PRIME) by a single operator. Measurements will be obtained from standard parasternal and apical views, according to the European Society of Cardiology recommendations.
  Left ventricular mass (g) will be estimated using the following formula:
  LV mass = 0.8 × {1.04 × [(LVEDD + PWTd + IVSd)³ - (LVEDD)³]} + 0.6 where: LVEDD = LV end-diastolic diameter PWTdP = posterior wall thickness in diastole IVSd = interventricular septal thickness in diastole
Gut Microbiota | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on the percentage change of the following measures relative to the baseline measures.
Systolic blood pressure | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on the percentage of the following measures relative to the baseline measures.
Diastolic blood pressure | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on the percentage of the following measures relative to the baseline measures.
Recovery of gestational weight gain | Visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on recovery of the gestational weight gain.
Glucose | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on the percentage change of the following measures relative to the baseline measures.
Haemoglobin A1c | Visit 1 (3rd trimester - 30-25 gestational weeks), visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of the dietary education counseling focused Mediterranean Diet promotion (intervention group) vs nutritional standard-care of the Portuguese National Health System (control group) on the percentage change of the following measures relative to the baseline measures.

OTHER OUTCOMES:
Age of Infant at Introduction of Complementary Feeding | Visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of dietary education counseling focused on Mediterranean Diet promotion (intervention group) vs nutritional standard care of the Portuguese National Health System (control group) on the timing of complementary feeding (solid food) introduction in infants.
  At every time points, mothers will be asked using structured parental questionnaires to report the infant's age (in weeks) at the introduction of any solid or semi-solid foods, excluding breast milk or infant formula.
  The primary metric will be the infant's age in weeks at first introduction of complementary feeding.
Duration of Exclusive Breastfeeding | Visit 2 (1 month postpartum), visit 3 (6 months postpartum) and visit 4 (12 months postpartum).
  To assess the effect of dietary education counseling focused on Mediterranean Diet promotion (intervention group) vs nutritional standard care of the Portuguese National Health System (control group) on the duration of exclusive breastfeeding.
  Exclusive breastfeeding is defined according to WHO criteria as providing only breast milk with no additional food or drink, not even water, except for oral rehydration solutions or drops/syrups of vitamins, minerals, or medicines.
  Data will be collected via structured parental. Mothers will report whether they are exclusively breastfeeding and the age (in weeks) at which exclusive breastfeeding stopped, if applicable.
  The outcome will be reported as the duration of exclusive breastfeeding in weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Inês Falcão Pires, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Unidade Local de Saúde de São João, Porto, Viana do Castelo District, Portugal